CLINICAL TRIAL: NCT05439460
Title: Management of Acute Pulmonary Hypertensive Crisis in Children With Known Pulmonary Arterial Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Chandra Ramamoorthy, Professor, Pediatric Cardiac Anesthesia, Stanford University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 22554
Record Dates: First submitted 2014-08-30; First posted 2022-06-30 (Actual); Results first posted 2022-08-05 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-07

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Phenylephrine; Epinephrine; Arginine Vasopressin; Vasopressins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Phenylephrine (Experimental): Phenylephrine will be administered once the child is under anesthesia and the interventional cardiologist has measured the pressures in the pulmonary artery.
  Interventions: Drug: Phenylephrine
- Epinephrine (Experimental): Epinephrine will be administered once the child is under anesthesia and the interventional cardiologist has measured the pressures in the pulmonary artery.
  Interventions: Drug: Epinephrine
- Arginine Vasopressin (Experimental): Arginine Vasopressin will be administered once the child is under anesthesia and the interventional cardiologist has measured the pressures in the pulmonary artery.
  Interventions: Drug: Arginine Vasopressin

INTERVENTIONS:
Drug: Phenylephrine — 5 subjects will get Phenylephrine during cardiac catheterization in patient with known Pulmonary Arterial Hypertension.Dose will be 1ug/kg body weight. Pressures in the pulmonary artery will be measured before and after the drug administration.
  Other Names: Phenylephrine Hydrochloride
  Arms: Phenylephrine
Drug: Epinephrine — 5 subjects will get Epinephrine during cardiac catheterization in patient with known Pulmonary Arterial Hypertension.Dose will be 0.5-1ug/kg body weight. Pressures in the pulmonary artery will be measured before and after the drug administration.
  Other Names: Epinephrine injection
  Arms: Epinephrine
Drug: Arginine Vasopressin — 5 subjects will get Arginine Vasopressin during cardiac catheterization in patient with known Pulmonary Arterial Hypertension.Dose will be 1ug/kg body weight. Pressures in the pulmonary artery will be measured before and after the drug administration.
  Other Names: Vasopressin injection
  Arms: Arginine Vasopressin

SUMMARY:
Pulmonary arterial hypertension (PAH) is a disease where the blood pressure in the pulmonary arteries (PAP) is high. PAH increases the risk of adverse events, including death, during and or after procedures. The severity of baseline PAH correlates with the incidence of major complications, such that those with PAP higher than their systemic blood pressure (SBP) had a 8 fold increased risk of complications. These children present for procedures where an acute exacerbation of their chronic illness-termed Pulmonary Hypertensive (PH)crisis, can occur, often resulting in death if not detected and managed expeditiously. Unfortunately there is little data and no consensus in the pediatric literature on how PH crisis should be managed.

--------------------------------------------------------------------------------

DETAILED DESCRIPTION:
Pulmonary arterial hypertension (PAH) is a disease where the blood pressure in the pulmonary arteries (PAP) is high. PAH increases the risk of adverse events, including death, during and or after procedures. The severity of baseline PAH correlates with the incidence of major complications, such that those with PAP higher than their systemic blood pressure (SBP) had a 8 fold increased risk of complications. These children present for procedures where an acute exacerbation of their chronic illness-termed PH crisis, can occur, often resulting in death if not detected and managed expeditiously. Unfortunately there is little data and no consensus in the pediatric literature on how PH crisis should be managed. Over the last 10 years we have developed considerable expertise in managing children with PAH and preventing and treating their acute crisis, using a medication called phenylephrine. This medication is routinely used to increase the blood pressure in patients (adults and children) to treat hypotension. Our theory has been that by increasing SBP, we can increase the blood flow to the coronary arteries and prevent the right ventricle from failing acutely. The latter results in catastrophic hypotension, heart arrythmias and death. There is no consensus or protocol guiding the management of the acute crisis. This purpose of this study is to close that gap.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting for cardiac catheterization procedure with a diagnosis of PAH either by previous cardiac catheterization or echocardiography

Exclusion Criteria:

* Children presenting for cardiac catheterization who do not have PAH;
* Children with PAH but with intracardiac shunts

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2012-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chandra Ramamoorthy, MD, Principal Investigator — Cardiac Anesthesia, Stanford University Medical Ctr.
Locations (1):
- Cardiac Catheterization Lab,Stanford University Medical Center, Stanford, California, United States

REFERENCES:
- [Background] Friesen RH, Williams GD. Anesthetic management of children with pulmonary arterial hypertension. Paediatr Anaesth. 2008 Mar;18(3):208-16. doi: 10.1111/j.1460-9592.2008.02419.x. PMID 18230063
- [Result] Siehr SL, Feinstein JA, Yang W, Peng LF, Ogawa MT, Ramamoorthy C. Hemodynamic Effects of Phenylephrine, Vasopressin, and Epinephrine in Children With Pulmonary Hypertension: A Pilot Study. Pediatr Crit Care Med. 2016 May;17(5):428-37. doi: 10.1097/PCC.0000000000000716. PMID 27144689

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were assigned sequentially; the first group received phenylephrine, the second group received arginine vasopressin, and the third group received epinephrine.
Groups:
- Phenylephrine: Phenylephrine (1ug/kg) administered once the child is under anesthesia.
- Arginine Vasopressin: Arginine Vasopressin (1ug/kg) administered once the child is under anesthesia.
- Epinephrine: Epinephrine (0.5-1ug/kg) administered once the child is under anesthesia.
Period: First Intervention (Approx 5h on Study)
Arm/Group | Phenylephrine | Arginine Vasopressin | Epinephrine
Started | 5 | 0 | 0
Completed | 5 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Second Intervention (Approx 5h on Study)
Arm/Group | Phenylephrine | Arginine Vasopressin | Epinephrine
Started | 0 | 5 | 0
Completed | 0 | 5 | 0
Not Completed | 0 | 0 | 0
Period: Third Intervention (Approx 5h on Study)
Arm/Group | Phenylephrine | Arginine Vasopressin | Epinephrine
Started | 0 | 0 | 5
Completed | 0 | 0 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phenylephrine | Arginine Vasopressin | Epinephrine | Total
Number analyzed (Participants) | 5 | 5 | 5 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.2 (3.8) | 10.5 (4.9) | 6.8 (4.2) | 9.2 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 3 | 11
  Male | 1 | 1 | 2 | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 5 | 5 | 15

OUTCOME MEASURES:

1. Primary Outcome: Change in Systemic Vascular Resistance Index (SVRI) to Pulmonary Vascular Resistance Index (PVRI) Ratio (Rp:Rs Ratio)
Description: In patients with pulmonary hypertension (PH) one anticipates a greater increase in pulmonary vascular resistance as opposed to systemic vascular resistance when vasopressors are administered.
Time Frame: Day 1 (at baseline and up to 5 minutes following study drug administration) (Q: 2 minutes - 2 to 5 minutes?)
Measure: Mean (Standard Deviation); unit: Rp:Rs ratio
Arm/Group | Phenylephrine | Arginine Vasopressin | Epinephrine
Number analyzed (Participants) | 5 | 5 | 5
Rp:Rs ratio
  Baseline | 0.8 (0.7) | 0.75 (0.41) | 0.61 (0.23)
  Approx. 2 minutes following drug administration | 0.73 (0.77) | 0.49 (0.24) | 0.6 (0.34)
Statistical Analysis 1: Comparison: Phenylephrine; Change in phenylephrine group; Test type: Other; p = 0.9, t-test, 2 sided
Statistical Analysis 2: Comparison: Arginine Vasopressin; Change in arginine vasopressin group; Test type: Other; p = 0.3, t-test, 2 sided — A p-value of <0.05 would be considered statistically significant
Statistical Analysis 3: Comparison: Epinephrine; Change in epinephrine group; Test type: Other; p = 1, t-test, 2 sided — A p-value of <0.05 would be considered statistically significant

ADVERSE EVENTS:
Time Frame: During procedure (approx. 5 h)
Arm/Group | Phenylephrine | Arginine Vasopressin | Epinephrine
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 2/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phenylephrine (N=5) | Arginine Vasopressin (N=5) | Epinephrine (N=5)
Transient arrhythmia (Cardiac disorders) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2011-11-08): https://cdn.clinicaltrials.gov/large-docs/60/NCT05439460/Prot_000.pdf
  • Statistical Analysis Plan (2016-05-01): https://cdn.clinicaltrials.gov/large-docs/60/NCT05439460/SAP_001.pdf